CLINICAL TRIAL: NCT03787082
Title: A Randomized Trial of Chlorhexidine Mouthwash and Oral Nitrate in Adults With Pulmonary Hypertension
Brief Title: Chlorhexidine Mouthwash and Oral Nitrate in Adults With Pulmonary Hypertension
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never able to start after the pandemic restrictions lifted
Sponsor: Gladwin, Mark, MD (Individual)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Alison Morris, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19120104; 5P01HL103455 (NIH)
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension; Heart Failure With Normal Ejection Fraction; Pulmonary Heart Disease and Diseases of Pulmonary Circulation
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Heart Disease | interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will receive open label nitrate and be randomly assigned to either chlorhexidine mouthwash or placebo mouthwash. The participant and investigator will be blinded to which mouthwash the participant is randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine Gluconate Mouthwash (Experimental): rinse with chlorhexidine gluconate 0.12% (15mL) mouthwash before administration of 14N Sodium Nitrate 1,000 mg/11.18 mmol, oral
  Interventions: Drug: Nitrates; Drug: Chlorhexidine Gluconate Mouthwash
- Placebo Mouthwash (Placebo Comparator): rinse with placebo mouthwash (15mL) before administration of 14N Sodium Nitrate 1,000 mg/11.18 mmol, oral
  Interventions: Drug: Nitrates; Drug: Placebo Mouthwash

INTERVENTIONS:
Drug: Nitrates — 1,000 mg/11.18 mmol, oral
  Other Names: 14N Sodium Nitrate
Drug: Chlorhexidine Gluconate Mouthwash — chlorhexidine gluconate 0.12% (15mL) mouth rinse for 1 minute
  Other Names: Chlorhexidine mouthwash
  Arms: Chlorhexidine Gluconate Mouthwash
Drug: Placebo Mouthwash — sterile water (15mL) mouth rinse for 1 minute
  Other Names: Sterile Water
  Arms: Placebo Mouthwash

SUMMARY:
This is an open-label, single-center study to examine distinguishing features of the structure and function of the oral and gut microbiome in volunteers with PH in the breakdown of oral nitrate and effect on hemodynamics.

DETAILED DESCRIPTION:
This is an open-label, single-center study to examine distinguishing features of the structure and function of the oral and gut microbiome in volunteers with PH in the breakdown of oral nitrate and effect on hemodynamics.

The investigators will enroll 40 PH patients over three years. 5 healthy participants will be enrolled as controls. Participants will receive a single dose of the study drug,:14N Sodium Nitrate(1000mg): standard sodium nitrate, and all will receive one dose of CLA 3g. CLA will be obtained from GNC (General Nutrition Corporation) and given once. Participants will be randomized to receive chlorhexidine gluconate 0.12% (15mL) or placebo to rinse their mouth with for 1 minute.

Oral samples will be collected pre- and post-chlorhexidine treatments and stool samples will be collected post-chlorhexidine treatment.

Right heart catheterization will be performed for clinical or research purposes.

The RHC done (in the last 5 years) that establishes inclusion is not the same RHC done as part of the study in most cases. If there is a strong suspicion of PH based on echocardiography in a patient who has not had a clinical RHC, the first hemodynamic measurements obtained in the clinical RHC will establish inclusion and the RHC study procedures will be performed following confirmation of inclusion.

Participants for whom the RHC done in the study is considered a clinical RHC will be participants who do have an additional follow up RHC scheduled.

Participants for whom the RHC done in the study is considered a research RHC will be those who do not have an additional follow RHC scheduled or who are considered healthy and have not had an RHC before.

Catheterization will generally be performed via the right internal jugular vein access with the assistance of fluoroscopy, if needed. Once the pulmonary arterial (PA) catheter has been placed in proper position, measured values will be obtained. The investigators often perform simultaneous measurement of right atrial pressure and distal pressure (PAP/PAWP) using two transducers in order to assess both pressures during vasodilator challenge, or other confrontational testing. An initial hemodynamic profile will be obtained.

With the right heart catheter still in place, participants will be randomized to either chlorhexidine mouthwash or placebo, then after 30 minutes, all will receive 14N oral nitrate and CLA. A repeat hemodynamic profile will be performed after two hours. Nitrate metabolites in plasma will be measured at time 0, 2, and 6 hrs after 14N nitrate dose. Urine nitrite and nitrate will be measured at 0 and 6 hours. Participants will be monitored with continuous pulse oximetry and EKG monitoring. Blood pressure measurements will be performed every 15 minutes during the catheterization. Pressure-volume loop and impedance analysis will be performed at the time of the right heart catheterization (RHC) using the micromanometer catheter technique to simultaneously measure RV pressure and pulmonary blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Undergoing clinical right heart catheterization or had a RHC in past 5 years if in PH group
* Pulmonary Hypertension: hemodynamically defined by a mean PAP ≥ 25 mm Hg and have a PVR > 3 Woods units and normal cardiac index (>2.0 L/min/m2)
* Healthy Control group: no history of or active cardiac or pulmonary disease
* Ability to provide written informed consent

Exclusion Criteria:

* Use of systemic antibiotics and/or chlorhexidine mouthwash within the previous three months
* Use of immune suppression (chemotherapy, oral prednisone greater than 20mg per day, etc) with in the previous three months
* Use of phosphodiesterase-5 inhibitors (tadalafil, sildenafil, etc) within 7 days before study drug administration
* Current pregnancy or lactation
* Uncontrolled systemic hypertension based on repeated measurement of sitting systolic blood pressure >185 mm Hg or sitting diastolic blood pressure >110 mm Hg
* Has chronic renal insufficiency as defined by serum creatinine >3 mg/dL in the last 6 months or requiring dialytic support as reported in the medical record
* Known history of left ventricular ejection fraction < 40% by multiple gated acquisition scan (MUGA), angiography, or echocardiography
* History of atrial septostomy
* Repaired or unrepaired congenital heart disease
* Pericardial constriction
* Restrictive or constrictive cardiomyopathy
* Symptomatic coronary disease with demonstrable ischemia
* Addition or change in dosing of hormonal contraception medications (OCP, IUD, Depo-Provera) in the past 4 weeks.
* Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study or would prevent completion of the study
* Active participation in other research studies with investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma Nitrate | At baseline and 2 hours post drug administration
Change in Urine Nitrate | At baseline and 2 hours post drug administration
Change in Plasma Nitrate | At baseline and 6 hours post drug administration
Change in Urine Nitrate | At baseline and 6 hours post drug administration
Change in Plasma Nitrate | At 2 hours post drug administration and 6 hours post drug administration
Change in Urine Nitrate | At 2 hours post drug administration and 6 hours post drug administration

SECONDARY OUTCOMES:
Change in Pulmonary Vascular Resistance (PVR) | At baseline and 2 hours post drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Alison Morris, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- Cathy Kessinger, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After de-identification, all participant data collected during the trial will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made following publication.
Access Criteria: Data will be available publicly.